CLINICAL TRIAL: NCT03192111
Title: A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Evaluate the Pharmacokinetics of Entinostat in Adult Subjects With Normal and Impaired Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics of Entinostat in Adult Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SNDX-275-0190
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Renal Impairment; Healthy Volunteer
Keywords: Healthy Volunteers; Mild Renal Impairment; Moderate Renal Impairment; Severe Renal Impairment; Entinostat; Histone Deacetylase Inhibitor; HDAC
MeSH Terms: conditions — Renal Insufficiency | interventions — entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild Renal Impairment (Experimental): Subjects with mild renal impairment
  Interventions: Drug: Entinostat
- Moderate Renal Impairment (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: Entinostat
- Severe Renal Impairment (Experimental): Subjects with severe renal impairment
  Interventions: Drug: Entinostat
- Healthy Subjects (Experimental): Healthy volunteers mean-matched to the mild, moderate, and severe renal impairment patients
  Interventions: Drug: Entinostat

INTERVENTIONS:
Drug: Entinostat — HDAC (histone deacetylase) inhibitor
  Other Names: SNDX-275; MS-275

SUMMARY:
This purpose of this study is to evaluate the effects of a single dose of entinostat on subjects with varying levels of renal impairment.

The primary objective of this study is to evaluate the pharmacokinetics of a single dose of entinostat in adult subjects with mild, moderate and severe renal impairment compared to healthy mean-matched subjects.

The secondary objective of this study is to evaluate the safety and tolerability of entinostat in adult subjects with mild, moderate, and severe renal impairment and in healthy mean-matched adult subjects.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. Adult male or female (of non childbearing potential only), at least 18 years of age, at screening.
2. BMI ≥ 18.5 to ≤ 40.0 kg/m2, at screening.
3. Subject is a non-smoker or moderate smoker (≤ 10 cigarettes/day or the equivalent). Subject must agree to consume no more than 10 cigarettes or equivalent/day from the time of screening and throughout the period of PK sample collection.
4. Females must be of non childbearing potential and must have undergone one of the following sterilization procedures, and have official documentation, at least 6 months prior to dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
5. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond dosing of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to dosing of study drug. A male who has been vasectomized less than 4 months prior to dosing must follow the same restrictions as a non vasectomized male).
6. If male, must agree not to donate sperm from dosing until 90 days after dosing of study drug.
7. Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

   Mild, Moderate, and Severe Renal Impaired Subjects:
8. Baseline health is judged to be stable based on medical history, laboratory profiles, vital signs, or ECGs at screening, as deemed by the PI. Subjects with any clinical laboratory results outside normal ranges may be enrolled if deemed appropriate in the opinion of the PI.
9. For subjects with mild RI only: Baseline eGFR 60 89 mL/min/1.73m2, inclusive, based on the MDRD equation at screening defined as follows:

   eGFR = 175 x (Scr,std)-1.154 x (Age)-0.203 Scr, std: serum creatinine (mg/dL) measured with a standardized assay. For females, multiply result by 0.742; if African American, multiply result by 1.212.

   For subjects with moderate RI only: Baseline eGFR 30 - 59 mL/min/1.73m2, inclusive, based on the MDRD equation at screening as described above.

   For subjects with severe RI only: Baseline eGFR 29 mL/min/1.73m2 or less based on the MDRD equation at screening as described above.
10. Subject has had no clinically significant change in renal status at least 1 month prior to study medication administration and is not currently or has not previously been on hemodialysis.

Matched Healthy Control Subjects 8. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. Subjects with any clinical laboratory results outside normal ranges may be enrolled if deemed appropriate in the opinion of the PI.

9. Has eGFR ≥ 90 mL/min/1.73m2, based on the MDRD equation at screening defined as follows: eGFR = 175 x (Scr,std)-1.154 x (Age)-0.203 Scr, std: serum creatinine (mg/dL) measured with a standardized assay. For females, multiply result by 0.742; if African American, multiply result by 1.212.

Actual creatinine clearance, as determined by a 24-hour urine collection, may be used in place of or in conjunction with the MDRD equation, at the PI's discretion. Subjects who have an actual or estimated creatinine clearance up to 10% below 90 mL/min/1.73m2 may be enrolled in the study at the discretion of the PI.

10. The age of individual healthy adult male and female subjects is aimed to be within the range of the mean age ± 10 years of the mild, moderate and severe RI subjects. In the event that these subjects do not match the mean for age in the severe RI cohort, additional healthy subjects (up to 8) will be enrolled using the same criteria.

11. The BMI of individual healthy adult male and female subjects is aimed to be within the range of the mean BMI ± 20 % of the mild, moderate and severe RI subjects. In the event that these subjects do not match the mean for BMI in the severe RI cohort, additional healthy subjects (up to 8) will be enrolled using the same criteria.

Exclusion Criteria:

All Subjects:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or drugs with a benzamide structure (e.g., tiapride, remoxipride, clebropride), related compounds, or inactive ingredients.
5. History or presence of any of the following as deemed clinically significant in the opinion of the PI or designee:
6. Cancer (subject with history of cancer that is in complete remission and not requiring treatment for at least 5 years, basal cell carcinoma or cervical intraepithelial neoplasia/cervical carcinoma in situ or melanoma in situ superficial skin lesions that have been successfully removed will not be exclusionary).
7. Active cardiovascular disorders (no history of myocardial infarction within 6 months of dosing, no stents or bypass within 6 months of dosing, ≥ Class 2 congestive heart failure).
8. Acute or chronic GI conditions (e.g., peptic ulcer, colitis, gastric bypass or equivalent) that would interfere with drug tolerance or absorption; subjects with cholecystectomy or uncomplicated gallbladder for over 1 year of dosing would be allowed.
9. Clinically significant infection within 1 month prior to dosing as determined by the PI or designee.
10. Female subjects of childbearing potential, pregnant or lactating subjects.
11. Positive results for the urine/saliva drug screen or for the urine/breath alcohol screen at screening or check-in unless the positive drug screen is due to prescription drug use and is approved by the PI and Sponsor.
12. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
13. Unable to refrain from or anticipates the use of:

    * Any drug known to be metabolized by CYP1A2 or CYP2C8, or to be a strong or moderate inhibitor of P gp or breast cancer resistance protein (BCRP) for 14 days prior to dosing and throughout the study. Use of weak inhibitors may be deemed acceptable following consultation with the Sponsor Medical Monitor and the PI. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamic interaction with study drug.
    * Any medication or substance (including prescription or over-the-counter, including herbal products, natural or herbal supplements) which cannot be discontinued at least 14 days prior to dosing and throughout the study. Subjects who are taking medications for stable diseases for at least ~2 weeks for subjects with severe RI or ~1 month for mild and moderate renal impaired subjects (or 5 half-lives of the compound, whichever is longer) prior to dosing will be allowed to participate in the study at the discretion of the PI and following consultation with the Sponsor Medical Monitor. See Section 10.4.2 for additional details on allowable and prohibited concomitant therapy.
14. Seated heart rate is equal to or lower than 40 bpm or higher than 99 bpm at screening.
15. Subject has had a renal transplant or has had nephrectomy.
16. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to dosing and throughout the study.
17. Donation of blood or significant blood loss within 56 days prior to dosing.
18. Plasma donation within 7 days prior to dosing.
19. Participation in another clinical study within 28 days prior to dosing. The 28 day window will be derived from the date of dosing.

    Mild, Moderate, and Severe Renal Impaired Subjects:
20. History or presence of alcoholism or drug abuse within the past 6 months prior to dosing.
21. Seated blood pressure is less than 90/40 mmHg or greater than 180/105 mmHg at screening.
22. PR interval > 240 msec, QRS > 140 msec at screening.
23. QTcF interval is >490 msec or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
24. Has rapidly fluctuating renal function as determined by historical measurements. Rapidly fluctuation renal function is defined as creatinine clearance that differs by more than 30% within 3 months of the screening eGFR determination. If historical measurements are not available, then the 2 measurements will be used to demonstrate stability.

Healthy Subjects:

20. History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.

21. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.

22. PR interval > 220 msec or QRS > 120 msec at screening. 23. QTcF interval is > 450 msec or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
To evaluate AUC0-t (area under the concentration-time curve) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  AUC0-t will be computed for all subjects
To evaluate AUC0-inf (area under the concentration-time curve, from time 0 to infinity) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  AUC0-inf will be computed for all subjects
To evaluate Cmax (maximum observed concentration) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  Cmax will be computed for all subjects

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (safety and tolerability) of entinostat in subjects with varying degrees of renal impairment and healthy mean-matched healthy subjects | Pre-dose to 14 days after last PK sample
  Subjects will be followed for adverse events up to 14 days after the last PK sample is collected.

OTHER OUTCOMES:
To evaluate AUC%extrap (percent of AUC0-inf extrapolated) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  AUC%extrap will be computed for all subjects
To evaluate Tmax (time to reach maximum observed concentration) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  Tmax will be computed for all subjects
To evaluate Kel (apparent terminal elimination rate constant) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  Kel will be computed for all subjects
To evaluate T 1/2 (apparent terminal elimination half-life) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  T 1/2 will be computed for all subjects
To evaluate CL/F (apparent total plasma clearance after oral [extravascular] administration) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects. | Pre-dose through Day 22
  CL/F will be computed for all subjects
To evaluate Vz/F (apparent volume of distribution during terminal elimination phase) for entinostat in subjects with varying degrees of renal impairment versus healthy matched subjects | Pre-dose through Day 22
  Vz/F will be computed for all subjects

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center for Clinical Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No